CLINICAL TRIAL: NCT05249829
Title: A Phase 2/3, Randomized, Observer-blind, Active-controlled, Multicenter Study to Evaluate the Immunogenicity and Safety of Omicron Variant Vaccines in Comparison With mRNA-1273 (Prototype) Booster Vaccine
Brief Title: A Study to Evaluate the Immunogenicity and Safety of Omicron Variant Vaccines in Comparison With mRNA-1273 Booster Vaccine for COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1273-P305; 2022-000063-51 (EudraCT Number)
Record Dates: First submitted 2022-02-19; First posted 2022-02-22 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: SARS-CoV-2
Keywords: Spikevax; mRNA-1273; mRNA-1273 vaccine; mRNA-1273.529; mRNA-1273.529 vaccine; Omicron; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna; Multivalent Vaccine; Variant Strains
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Phase A of this study will be observer-blinded. Phase B of the study will be open-label and blinding is not applicable
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: mRNA-1273.529 (Experimental): Phase A: Participants will receive 1 intramuscular (IM) dose of mRNA-1273.529 on Day 1.
  Phase B: After Day 179, eligible participants may choose to be unblinded and to receive an additional booster outside of the study.
  Interventions: Biological: mRNA-1273.529
- Part 1: mRNA-1273 (Active Comparator): Phase A: Participants will receive 1 IM dose of mRNA-1273 on Day 1.
  Phase B: After Day 179, eligible participants may choose to be unblinded and to receive an additional booster outside of the study.
  Interventions: Biological: mRNA-1273
- Part 2: mRNA-1273.214 (Experimental): Phase A: Participants will receive 1 IM dose of mRNA-1273.214 on Day 1.
  Phase B: After Day 85, eligible participants may choose to be unblinded and to receive an additional booster outside of the study.
  Interventions: Biological: mRNA-1273.214
- Part 2: mRNA-1273 (Active Comparator): Phase A: Participants will receive 1 IM dose of mRNA-1273 on Day 1.
  Phase B: After Day 85, eligible participants may choose to be unblinded and to receive an additional booster outside of the study.
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: mRNA-1273.529 — Sterile liquid for injection
  Arms: Part 1: mRNA-1273.529
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: Part 1: mRNA-1273; Part 2: mRNA-1273
Biological: mRNA-1273.214 — Sterile liquid for injection
  Arms: Part 2: mRNA-1273.214

SUMMARY:
This is a 2-part study to evaluate the immunogenicity, safety, and reactogenicity of mRNA-1273.529 and mRNA-1273.214 administered as a booster dose.

DETAILED DESCRIPTION:
In Part 1, participants will be randomized in a 1:1 ratio to receive a single dose of either mRNA-1273.529 or mRNA-1273.

In Part 2, participants will be randomized in a 1:1 ratio to receive a single dose of either mRNA-1273.214 or mRNA-1273.

All participants will have previously received 2 or 3 doses of an authorized/approved COVID-19 vaccine. Participants who previously received 2 doses of a COVID-19 vaccine as a primary series will receive mRNA-1273.529, mRNA-1273.214, or mRNA-1273 as the 3rd dose, and participants who have previously received a primary series and 1 booster dose will receive mRNA-1273.529, mRNA-1273.214, or mRNA-1273 as the 4th dose (a mixed approach is acceptable). Each part will include Phase A (randomized, blinded) and Phase B (open-label, observational).

ELIGIBILITY:
Inclusion Criteria:

* Female participants of childbearing potential may be enrolled in the study if the participant has a negative pregnancy test at the Screening Visit and on the day of vaccination prior to vaccine dose being administered on Day 1; has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose (Day 1); and has agreed to continue adequate contraception through 90 days following vaccine administration.
* Participant has received 2 prior doses of one of the following approved/authorized COVID-19 vaccines: Moderna, Pfizer/BioNTech, Oxford/AstraZeneca, Janssen. A heterologous vaccine regimen is acceptable.
* Participants who will receive the 4th dose as part of the study must have previously received a mRNA vaccine (Moderna or Pfizer/BioNTech) as the 3rd dose of a COVID-19 vaccine. Participants who will receive the 3rd dose as part of the study may have previously received 2 doses of an approved/authorized mRNA or a non-mRNA COVID-19 vaccine (a heterologous vaccine regimen is acceptable).

Exclusion Criteria:

* Participant had close contact (without personal protective equipment [PPE]) as defined by the Centers for Disease Control and Prevention (CDC) in the past 14 days to someone diagnosed with SARS-CoV-2 infection or COVID-19 within 10 days of the close contact. Participants may be rescreened after 14 days provided that they remain asymptomatic.
* Participant is acutely ill or febrile (temperature ≥ 38.0°C/100.4°F) 72 hours prior to or at the Screening Visit or Day 1.
* Participant has tested positive for SARS-CoV-2 by an authorized/approved lateral flow/rapid antigen or polymerase chain reaction (PCR) test within 90 days of Screening.
* Participant has received a COVID-19 vaccine within 90 days of the Screening Visit.
* Participant has received a total of 4 doses or more of COVID-19 vaccine.
* Participant has received a COVID-19 vaccine at a dose different from the authorized/approved dose.
* Any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 181 days prior to screening (for corticosteroids ≥10 milligrams [mg]/day of prednisone or equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Participant has received or plans to receive any licensed vaccine ≤28 days prior to the study injection (Day 1) or plans to receive a licensed vaccine within 28 days after the study injection (with the exception that approved seasonal influenza vaccine may be received by at least 7 days and preferably 14 days apart from the study injection).
* Participant has received systemic immunoglobulins or blood products within 90 days prior to the Screening Visit or plans to receive during the study.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.
* Participant has participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3548 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United Kingdom (29):
  - Aberdeen Royal Infirmary - PPDS, Aberdeen, Aberdeenshire
  - Southmead Hospital, Bristol, Avon
  - Wansford and Kingscliffe Practice, Wansford, Cambridgeshire
  - Halton General Hospital, Runcorn, Cheshire
  - The James Cook University Hospital, Middlesbrough, Cleveland
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Gloucester Royal Hospital, Gloucester, Gloucestershire
  - Portsmouth Research Hub, Portsmouth, Hampshire
  - Fylde Coast Clinical Research, Blackpool, Lancashire
  - Leicester General Hospital, Leicester, Leicestershire
  - Salford Royal Hospital - PPDS, Salford, Manchester
  - University College London Hospitals Covid-19 Vaccine Centre, London, Middlesex
  - Castle Hill Hospital, Hull, North Humberside
  - The Princess Royal Hospital, Telford, Shropshire
  - Royal United Hospital, Bath, Somerset
  - Sheffield/Northern General Hospital, Sheffield, South Yorkshire
  - Royal Glamorgan Hospital - PPDS, Pont-y-clun, Wales
  - Bradford Institute for Health Research, Bradford, West Yorkshire
  - Great Western Hospital, Swindon, Wiltshire
  - Queen Elizabeth Hospital, Birmingham
  - Barts Hospital, London
  - Royal Free Hospital, London
  - Kings College Hospital, London
  - Chelsea and Westminster Hospital, London
  - St. George's Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee IT, Cosgrove CA, Moore P, Bethune C, Nally R, Bula M, Kalra PA, Clark R, Dargan PI, Boffito M, Sheridan R, Moran E, Darton TC, Burns F, Saralaya D, Duncan CJA, Lillie PJ, San Francisco Ramos A, Galiza EP, Heath PT, Girard B, Parker C, Rust D, Mehta S, de Windt E, Sutherland A, Tomassini JE, Dutko FJ, Chalkias S, Deng W, Chen X, Feng J, Tracy L, Zhou H, Miller JM, Das R; Study Investigators. Omicron BA.1-containing mRNA-1273 boosters compared with the original COVID-19 vaccine in the UK: a randomised, observer-blind, active-controlled trial. Lancet Infect Dis. 2023 Sep;23(9):1007-1019. doi: 10.1016/S1473-3099(23)00295-5. Epub 2023 Jun 19. PMID 37348519

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 3779 participants who were screened for Part 1 and Part 2 of the study, 220 participants failed screening and 11 did not receive study vaccine.
Groups:
- Part 1: mRNA-1273.529: Phase A: Participants received 1 intramuscular (IM) dose of mRNA-1273.529 on Day 1. Phase B: After Day 179, eligible participants were allowed to choose to be unblinded and to receive an additional booster outside of the study.
- Part 1: mRNA-1273: Phase A: Participants received 1 IM dose of mRNA-1273 on Day 1. Phase B: After Day 179, eligible participants were allowed to choose to be unblinded and to receive an additional booster outside of the study.
- Part 2: mRNA-1273.214: Phase A: Participants received 1 IM dose of mRNA-1273.214 on Day 1. Phase B: After Day 85, eligible participants were allowed to choose to be unblinded and to receive an additional booster outside of the study.
- Part 2: mRNA-1273: Phase A: Participants received 1 IM dose of mRNA-1273 on Day 1. Phase B: After Day 85, eligible participants were allowed to choose to be unblinded and to receive an additional booster outside of the study.
Period: Overall Study
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Started | 367 | 357 | 1422 | 1402
Received at Least 1 Dose of Study Drug | 367 (Safety Set) | 357 (Safety Set) | 1422 (Safety Set) | 1402 (Safety Set)
Completed | 337 | 320 | 1314 | 1295
Not Completed | 30 | 37 | 108 | 107
Not completed — Participant Relocation | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 17 | 40 | 35
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 16 | 57 | 60
Not completed — Adverse Event | 2 | 2 | 2 | 2
Not completed — COVID-19 Non-Infection Related | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 5 | 3
Not completed — Death | 0 | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Safety Set included all randomized participants who received the study vaccine. Participants were included in the study vaccine arm that they actually received.
Groups:
- Part 1: mRNA-1273.529: Phase A: Participants received 1 IM dose of mRNA-1273.529 on Day 1. Phase B: After Day 179, eligible participants were allowed to choose to be unblinded to receive an additional booster outside of the study.
- Part 1: mRNA-1273: Phase A: Participants received 1 IM dose of mRNA-1273 on Day 1. Phase B: After Day 179, eligible participants were allowed to choose to unblinded to receive an additional booster outside of the study.
- Part 2: mRNA-1273.214: Phase A: Participants received 1 IM dose of mRNA-1273.214 on Day 1. Phase B: After Day 85, eligible participants were allowed to choose to be unblinded to receive an additional booster outside of the study.
- Part 2: mRNA-1273: Phase A: Participants received 1 IM dose of mRNA-1273 on Day 1. Phase B: After Day 85, eligible participants were allowed to choose to be unblinded and receive an additional booster outside of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273 | Total
Number analyzed (Participants) | 367 | 357 | 1422 | 1402 | 3548
Age, Customized [Number; unit: participants]
  >=16 and <65 Years | 241 | 235 | 945 | 935 | 2356
  >=65 Years | 126 | 122 | 477 | 467 | 1192
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 202 | 695 | 694 | 1791
  Male | 167 | 155 | 727 | 708 | 1757
Race/Ethnicity, Customized [Number; unit: participants]
  White | 353 | 335 | 1347 | 1313 | 3348
  Mixed or Multiple Ethnic Groups | 3 | 5 | 21 | 27 | 56
  Asian or Asian British | 10 | 10 | 31 | 41 | 92
  Black, African, Caribbean, or Black British | 0 | 0 | 6 | 6 | 12
  Other Ethnic Group | 1 | 5 | 4 | 7 | 17
  Not Reported | 0 | 2 | 11 | 7 | 20
  Unknown | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Geometric Mean Concentration (GMC) of mRNA-1273.529 and mRNA-1273 Against the B.1.1.529 Strain at Day 29
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. Results are reported as absorbance units/millilitre (AU/mL). The GMC 95% confidence interval (CI) was calculated based on the t-distribution of the log-transformed values then back-transformed to the original scale for presentation.
Time Frame: Day 29 (post vaccination)
Population: Per-Protocol Set for Immunogenicity-SARS-CoV-2 negative (PPSI-Neg) included all randomized participants who received the planned dose of study vaccine, had no major protocol deviations with an impact on critical or key study data, and had no serologic or virologic evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection at Baseline and up to the analysis visit. Here, Number of Participants Analysed: those participants who were evaluable for this Outcome Measure.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273
Number analyzed (Participants) | 274 | 277
AU/mL | 537.7 (478.2) [478.2 to 604.6] | 302.8 (274.8) [274.8 to 333.6]
Statistical Analysis 1: Comparison: Part 1: mRNA-1273.529 vs Part 1: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.529/GMCmRNA-1273 against the B.1.1.529 strain at Day 29 after study vaccine administration; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >0.667; Geometric Mean Ratio = 1.730, 99% CI 2-sided [1.493 to 2.005]

2. Primary Outcome: Part 1: GMC of mRNA-1273.529 and mRNA-1273 Against the B.1.1.529 Strain at Day 85
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. Results are reported as AU/mL. The GMC 95% CI was calculated based on the t-distribution of the log-transformed values then back-transformed to the original scale for presentation.
Time Frame: Day 85 (post vaccination)
Population: PPSI-Neg included all randomized participants who received the planned dose of study vaccine, had no major protocol deviations with an impact on critical or key study data, and had no serologic or virologic evidence of SARS-CoV-2 infection at Baseline and up to the analysis visit. Here, Number of Participants Analysed signifies those participants who were evaluable for this Outcome Measure.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273
Number analyzed (Participants) | 234 | 226
AU/mL | 284.7 (248.0) [248.0 to 326.7] | 152.6 (135.1) [135.1 to 172.3]
Statistical Analysis 1: Comparison: Part 1: mRNA-1273.529 vs Part 1: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.529/GMCmRNA-1273 against the B.1.1.529 strain at Day 85 after study vaccine administration; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower bound of the 96% CI of the Geometric Mean Ratio was >0.667; Geometric Mean Ratio = 1.763, 96% CI 2-sided [1.546 to 2.010]

3. Primary Outcome: Part 2: GMC of mRNA-1273.214 and mRNA-1273 Against the B1.1.529 Strain at Day 29
Description: as for outcome 2
Time Frame: Day 29 (post vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 968 | 894
AU/mL | 465.7 (437.0) [437.0 to 496.3] | 311.0 (292.9) [292.9 to 330.1]
Statistical Analysis 1: Comparison: Part 2: mRNA-1273.214 vs Part 2: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.214/GMCmRNA-1273 against the B.1.1.529 strain at Day 29 after study vaccine administration; Test type: Other — Non-inferiority was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >0.667. Superiority was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >1; Geometric Mean Ratio = 1.535, 99% CI 2-sided [1.409 to 1.672]

4. Primary Outcome: Part 2: GMC of mRNA-1273.214 and mRNA-1273 Against the B1.1.529 Strain at Day 85
Description: as for outcome 2
Time Frame: Day 85 (post vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 761 | 688
AU/mL | 258.2 (239.3) [239.3 to 278.7] | 153.0 (142.2) [142.2 to 164.6]
Statistical Analysis 1: Comparison: Part 2: mRNA-1273.214 vs Part 2: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.214/GMCmRNA-1273 against the B.1.1.529 strain at Day 85 after study vaccine administration; Test type: Other — [test comment as in outcome 3, analysis 1]; Geometric Mean Ratio = 1.713, 96% CI 2-sided [1.583 to 1.853]

5. Primary Outcome: Part 2: GMC of mRNA-1273.214 and mRNA-1273 Against the Ancestral Strain at Day 29
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. The ancestral (prototype) strain was Wuhan-Hu-1. Results are reported as AU/mL. The GMC 95% CI was calculated based on the t-distribution of the log-transformed values then back-transformed to the original scale for presentation.
Time Frame: Day 29 (post vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 951 | 880
AU/mL | 2998.8 (2825.4) [2825.4 to 3182.8] | 2933.6 (2772.3) [2772.3 to 3104.4]
Statistical Analysis 1: Comparison: Part 2: mRNA-1273.214 vs Part 2: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.214/GMCmRNA-1273 against the ancestral strain at Day 29 after study vaccine administration. Reported statistical analysis based upon the number of participants with non-missing data at baseline and the corresponding timepoint (N=1818); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >0.667; Geometric Mean Ratio = 1.048, 99% CI 2-sided [0.958 to 1.147]

6. Primary Outcome: Part 2: GMC of mRNA-1273.214 and mRNA-1273 Against the Ancestral Strain ay Day 85
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. The ancestral strain was Wuhan-Hu-1. Results are reported as AU/mL. The GMC 95% CI was calculated based on the t-distribution of the log-transformed values then back-transformed to the original scale for presentation.
Time Frame: Day 85 (post vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 761 | 685
AU/mL | 1753.1 (1650.0) [1650.0 to 1862.6] | 1610.2 (1519.6) [1519.6 to 1706.2]
Statistical Analysis 1: Comparison: Part 2: mRNA-1273.214 vs Part 2: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.214/GMCmRNA-1273 against the ancestral strain at Day 85 after study vaccine administration. Reported statistical analysis based upon the number of participants with non-missing data at baseline and the corresponding timepoint (N=1418); Test type: Other — Non-inferiority was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >0.667; Geometric Mean Ratio = 1.104, 96% CI 2-sided [1.032 to 1.180]

7. Primary Outcome: Parts 1 and 2: Percentage of Participants With Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs)
Description: Reactogenicity refers to the occurrence and intensity of selected signs and symptoms (ARs) occurring after vaccine injection. Participants recorded such occurrences in an electronic diary on the day of study vaccine injection and for the 7 days after the day of dosing. Solicited local ARs were injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of the injection. Solicited systemic ARs were headache, fatigue, myalgia (muscle aches all over the body), arthralgia (joint aches in several joints), nausea/vomiting, chills, and fever (oral temperature). The Investigator determined if a solicited AR was also to be recorded as an adverse event (AE). A summary of all Serious and Non Serious AEs, regardless of causality, is located in the 'Adverse Events' section.
Time Frame: Up to Day 8 (7 days post-vaccination)
Population: The Solicited Safety Set included all randomized participants who received the study vaccine and contributed any solicited AR data within the first 7 days after study vaccine administration. Participants were included in the study vaccine arm that they actually received. Here, Overall number of Participants Analyzed signifies those participants who were evaluable for this Outcome Measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 367 | 357 | 1421 | 1398
percentage of participants
  Any Solicited Local ARs | 84.5 (80.4) [80.4 to 88.0] | 89.1 (85.4) [85.4 to 92.1] | 83.6 (81.6) [81.6 to 85.5] | 89.9 (88.2) [88.2 to 91.4]
  Any Solicited Systemic ARs | 69.8 (64.8) [64.8 to 74.4] | 74.2 (69.4) [69.4 to 78.7] | 70.2 (67.7) [67.7 to 72.5] | 75.3 (73.0) [73.0 to 77.6]

8. Primary Outcome: Parts 1 and 2: Number of Participants With Unsolicited AEs
Description: An AE was any untoward medical occurrence associated with the use of a drug/vaccine, whether or not considered related to the drug/vaccine. An unsolicited AE was any AE reported by the participant that was not specified as a solicited AR in the protocol or was specified as a solicited AR but starts outside the protocol-defined period for reporting solicited ARs (that is, 7 days after vaccination). A summary of all Serious and Non Serious AEs, regardless of causality, is located in the 'Adverse Events' section.
Time Frame: Up to Day 29 (28 days post-vaccination)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 367 | 357 | 1422 | 1402
Participants | 142 | 124 | 442 | 429

9. Primary Outcome: Parts 1 and 2: Number of Participants With Serious AEs (SAEs)
Description: An AE was considered an SAE if, in the view of either the investigator or Sponsor, it resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization (hospitalization or prolongation of hospitalization in the absence of a precipitating event was not in itself an SAE), resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, was a congenital anomaly/birth defect, or was a medically important event. A summary of all Serious and Non Serious AEs, regardless of causality, is located in the 'Adverse Events' section.
Time Frame: Day 1 to end of study (Day 359)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 367 | 357 | 1422 | 1402
Participants | 20 | 13 | 60 | 72

10. Primary Outcome: Parts 1 and 2: Number of Participants With Medically Attended AEs (MAAEs)
Description: An MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner (HCP). This would include visits to a clinic for unscheduled assessments (for example, rash assessment, abnormal laboratory follow-up, coronavirus disease 2019 [COVID-19]) and visits to HCPs external to the clinic (for example, urgent care, primary care physician). A summary of all Serious and Non Serious AEs, regardless of causality, is located in the 'Adverse Events' section.
Time Frame: Day 1 to end of study (Day 359)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 367 | 357 | 1422 | 1402
Participants | 242 | 257 | 956 | 964

11. Primary Outcome: Parts 1 and 2: Number of Participants With AEs Leading to Withdrawal
Description: An AE leading to withdrawal was defined as any AE that caused the participant to withdraw from the study, regardless of whether the decision to withdraw from the study was made by the participant or by the Investigator. A summary of all Serious and Non Serious AEs, regardless of causality, is located in the 'Adverse Events' section.
Time Frame: Day 1 to end of study (Day 359)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 367 | 357 | 1422 | 1402
Participants | 2 | 3 | 3 | 6

12. Primary Outcome: Parts 1 and 2: Number of Participants With AEs of Special Interest (AESIs)
Description: An AESI is an AE (serious or non serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the investigator to the Sponsor was required. Such events may have required further investigation to characterize and understand them. A summary of all Serious and Non Serious AEs, regardless of causality, is located in the 'Adverse Events' section.
Time Frame: Day 1 to end of study (Day 359)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 367 | 357 | 1422 | 1402
Participants | 42 | 28 | 60 | 60

13. Secondary Outcome: Part 1: GMC of mRNA-1273.529 and mRNA-1273 Against the B.1.1.529 Strain at Day 29 and Day 85
Description: Blood samples for immunogenicity assessments were collected during protocol specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. Results are reported as AU/mL. The GMC 95% CI was calculated based on the t-distribution of the log-transformed values then back transformed to the original scale for presentation. Superiority at Day 29 was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >1. Superiority at Day 85 was demonstrated if the lower bound of the 96% CI of the Geometric Mean Ratio was >1.
Time Frame: Day 29 and Day 85 (post vaccination)
Population: PPSI-Neg included all randomized participants who received the planned dose of study vaccine, had no major protocol deviations with an impact on critical or key study data, and had no serologic or virologic evidence of SARS-CoV-2 infection at Baseline and up to the analysis visit. Here, Overall Number of Participants Analyzed signifies those participants who were evaluable for this Outcome Measure. Number Analyzed signifies those participants who were evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273
Number analyzed (Participants) | 274 | 277
AU/mL
  Day 29 | 537.7 [478.2 to 604.6] | 302.8 [274.8 to 333.6]
  Day 85: number analyzed (Participants) | 234 | 226
  Day 85 | 284.7 [248.0 to 326.7] | 152.6 [135.1 to 172.3]
Statistical Analysis 1: Comparison: Part 1: mRNA-1273.529 vs Part 1: mRNA-1273; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority was demonstrated if the lower bound of the 99% CI of the Geometric Mean Ratio was >1; Geometric Mean Ratio = 1.730, 99% CI 2-sided [1.493 to 2.005]
Statistical Analysis 2: Comparison: Part 1: mRNA-1273.529 vs Part 1: mRNA-1273; Geometric Mean Ratio = GMCmRNA-1273.529/GMCmRNA-1273 against the B.1.1.529 strain at Day 85 after study vaccine administration. Reported statistical analysis based upon the number of participants with non-missing data at baseline and the corresponding timepoint (N=460); Test type: Superiority — Superiority was demonstrated if the lower bound of the 96% CI of the Geometric Mean Ratio was >1; Geometric Mean Ratio = 1.763, 96% CI 2-sided [1.546 to 2.010]

14. Secondary Outcome: Part 1: GMC of mRNA-1273.529 and mRNA-1273 Against the B.1.1.529 Strain at Day 179
Description: Blood samples for immunogenicity assessments were collected during protocol specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. Results are reported as AU/mL. The GMC 95% CI was calculated based on the t-distribution of the log-transformed values then back transformed to the original scale for presentation.
Time Frame: Day 179 (post vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273
Number analyzed (Participants) | 160 | 138
AU/mL | 144.3 (119.4) [119.4 to 174.5] | 70.1 (59.0) [59.0 to 83.4]

15. Secondary Outcome: Part 1: GMC of mRNA-1273.529 and mRNA-1273 Against the Ancestral Strain at Day 29, Day 85, and Day 179
Description: as for outcome 6
Time Frame: Day 29, Day 85, Day 179 (post vaccination)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273
Number analyzed (Participants) | 270 | 272
AU/mL
  Day 29 | 2699.7 [2431.3 to 2997.7] | 3020.6 [2776.5 to 3286.2]
  Day 85: number analyzed (Participants) | 234 | 226
  Day 85 | 1401.2 [1236.9 to 1587.4] | 1559.4 [1401.2 to 1735.5]
  Day 179: number analyzed (Participants) | 160 | 133
  Day 179 | 734.6 [621.8 to 867.9] | 747.6 [644.1 to 867.7]

16. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Seroresponse Against SARS-CoV-2
Description: Seroresponse was defined by an increase of the GMC from pre-study vaccination (booster) below the lower limit of quantitation (LLOQ) to at least 4×LLOQ, or a 4-fold or greater rise if pre-study vaccination was ≥LLOQ. The number of participants analysed from the PPSI-Neg population include those with non-missing data at Baseline and the corresponding timepoint. 95% CI calculated using the Clopper-Pearson method.
Time Frame: Days 29, 85, 179, and 359
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 274 | 277 | 968 | 894
percentage of participants
  Day 29 - B.1.1.529 Strain | 83.2 [78.2 to 87.4] | 55.2 [49.2 to 61.2] | 84.7 [82.3 to 86.9] | 70.4 [67.2 to 73.3]
  Day 85 - B.1.1.529 Strain: number analyzed (Participants) | 234 | 226 | 761 | 688
  Day 85 - B.1.1.529 Strain | 48.3 [41.7 to 54.9] | 15.9 [11.4 to 21.4] | 60.6 [57.0 to 64.1] | 32.3 [28.8 to 35.9]
  Day 179 - B.1.1.529 Strain: number analyzed (Participants) | 160 | 138 | 546 | 507
  Day 179 - B.1.1.529 Strain | 18.1 [12.5 to 25.0] | 2.9 [0.8 to 7.3] | 37.5 [33.5 to 41.8] | 25.8 [22.1 to 29.9]
  Day 359 - B.1.1.529 Strain: number analyzed (Participants) | 74 | 61 | 286 | 251
  Day 359 - B.1.1.529 Strain | 36.5 [25.6 to 48.5] | 26.2 [15.8 to 39.1] | 32.5 [27.1 to 38.3] | 25.1 [19.9 to 30.9]
  Day 29 - Ancestral Strain: number analyzed (Participants) | 267 | 271 | 945 | 873
  Day 29 - Ancestral Strain | 43.1 [37.1 to 49.2] | 59.0 [52.9 to 65.0] | 70.9 [67.9 to 73.8] | 68.4 [65.2 to 71.5]
  Day 85 - Ancestral Strain: number analyzed (Participants) | 231 | 225 | 747 | 671
  Day 85 - Ancestral Strain | 14.3 [10.0 to 19.5] | 21.8 [16.6 to 27.7] | 38.8 [35.3 to 42.4] | 33.4 [29.8 to 37.1]
  Day 179 - Ancestral Strain: number analyzed (Participants) | 158 | 132 | 531 | 487
  Day 179 - Ancestral Strain | 2.5 [0.7 to 6.4] | 6.1 [2.7 to 11.6] | 25.0 [21.4 to 29.0] | 23.8 [20.1 to 27.9]
  Day 359 - Ancestral Strain: number analyzed (Participants) | 73 | 61 | 280 | 247
  Day 359 - Ancestral Strain | 2.7 [0.3 to 9.5] | 8.2 [2.7 to 18.1] | 8.9 [5.9 to 12.9] | 12.6 [8.7 to 17.3]

17. Secondary Outcome: Part 2: GMC of mRNA-1273.214 and mRNA-1273 Against Other Variant Strains
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody levels were measured by pseudovirus neutralization assays. Results are reported as AU/mL. The GMC 95% CI was calculated based on the t-distribution of the log-transformed values then back-transformed to the original scale for presentation. Other variant strains include B.1.1.7 Strain, AY.4 Strain, P.1 Strain.
Time Frame: Days 29 and 85
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 968 | 895
AU/mL
  Day 29 - B.1.1.7 Strain | 236533.1 [227116.7 to 246340.0] | 225834.1 [216536.7 to 235530.8]
  Day 85 - B.1.1.7 Strain: number analyzed (Participants) | 761 | 688
  Day 85 - B.1.1.7 Strain | 133951.9 [127594.4 to 140626.1] | 124778.3 [118785.1 to 131073.9]
  Day 29 - AY.4 Strain | 244715.5 [234951.9 to 254884.8] | 236066.3 [226310.8 to 246242.3]
  Day 85 - AY.4 Strain: number analyzed (Participants) | 761 | 688
  Day 85 - AY.4 Strain | 134119.3 [127672.7 to 140891.4] | 127263.6 [121106.4 to 133733.8]
  Day 29 - P.1 Strain | 182396.9 [175235 to 189850.9] | 175216.7 [168018.0 to 182723.9]
  Day 85 - P.1 Strain: number analyzed (Participants) | 761 | 688
  Day 85 - P.1 Strain | 103438.9 [98607.6 to 108506.8] | 97927.0 [93264.0 to 102823.2]

18. Secondary Outcome: Part 2: Percentage of Participants With Asymptomatic SARS-CoV-2 Infection Measured by Reverse Transcriptase Polymerase-chain Reaction (RT-PCR)
Description: Asymptomatic SARS-CoV-2 infection was defined as a positive RT-PCR test on a respiratory sample in the absence of symptoms or a positive serologic test for antinucleocapsid antibody after a negative test at time of enrollment.
Time Frame: Day 14 through the end of study (Day 359)
Population: Per-Protocol Set for Efficacy included all participants with a pre-vaccination/Baseline SARS-CoV-2 negative status who received the planned dose of study vaccination and had no major protocol deviations that had an impact on key or critical data.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 995 | 932
percentage of participants | 16.9 | 17.7

19. Secondary Outcome: Part 2: Percentage of Participants With Symptomatic SARS-CoV-2 Infection Measured by RT-PCR
Description: Symptomatic SARS-CoV-2 infection was defined 2 ways: protocol-defined COVID-19 and Center for Disease Control (CDC) COVID-19. Protocol-defined COVID-19 required at least 2 of the following systemic symptoms: fever, chills, myalgia, headache, sore throat, new olfactory and taste disorder(s), or at least 1 of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, or clinical/radiographical evidence of pneumonia, and at least 1 positive nasopharyngeal swab, nasal swab, or saliva sample (RT-PCR). CDC-defined COVID-19 was based on a positive respiratory sample (RT-PCR) and at least 1 of the following systemic or respiratory symptoms: fever, chills, cough, shortness of breath, and/or difficulty breathing, fatigue, muscle and/or body aches, headache, new loss of taste/smell, sore throat, congestion, runny nose, nausea, vomiting, or diarrhoea.
Time Frame: Day 1 through the end of study (Day 359)
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 995 | 932
percentage of participants | 50.8 | 48.6

20. Secondary Outcome: Part 2: Percentage of Participants With Primary Case Definition of COVID-19
Description: The primary case definition of COVID-19 (protocol-defined COVID-19) required the participant to have experienced at least 2 of the following systemic symptoms: fever, chills, myalgia, headache, sore throat, new olfactory and taste disorder(s), or the participant must have experienced at least 1 of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, or clinical or radiographical evidence of pneumonia, and must have at least 1 nasopharyngeal swab, nasal swab, or saliva sample (or respiratory sample, if hospitalized) positive for SARS-CoV-2 by RT-PCR.
Time Frame: Day 14 through the end of study (Day 359)
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 995 | 932
percentage of participants | 30.5 | 29.1

21. Secondary Outcome: Part 2: Percentage of Participants With Secondary Case Definition of COVID-19
Description: The secondary case definition of COVID-19 (CDC case definition) was based on a positive RT-PCR test on a respiratory sample and at least 1 of the following systemic or respiratory symptoms: fever, chills, cough, shortness of breath, and/or difficulty breathing, fatigue, muscle and/or body aches (not related to exercise), headache, new loss of taste/smell, sore throat, congestion, runny nose, nausea, vomiting, or diarrhoea.
Time Frame: Day 14 through the end of study (Day 359)
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
Number analyzed (Participants) | 995 | 932
percentage of participants | 33.5 | 30.9

ADVERSE EVENTS:
Time Frame: Day 1 to end of study (Day 359)
Description: The Safety Set included all randomized participants who received the study vaccine. Note, not all solicited ARs were considered AEs. Investigator determined if solicited AR was also to be recorded as an AE.
Arm/Group | Part 1: mRNA-1273.529 | Part 1: mRNA-1273 | Part 2: mRNA-1273.214 | Part 2: mRNA-1273
All-Cause Mortality (participants affected / at risk) | 0/367 | 1/357 | 2/1422 | 4/1402
Serious Adverse Events (participants affected / at risk) | 20/367 | 13/357 | 60/1422 | 72/1402
Other Adverse Events (participants affected / at risk) | 68/367 | 70/357 | 207/1422 | 198/1402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: mRNA-1273.529 (N=367) | Part 1: mRNA-1273 (N=357) | Part 2: mRNA-1273.214 (N=1422) | Part 2: mRNA-1273 (N=1402)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right aortic arch (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Richter's hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
High-grade B- cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (2)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motor neurone disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oromandibular dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Idiopathic angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: mRNA-1273.529 (N=367) | Part 1: mRNA-1273 (N=357) | Part 2: mRNA-1273.214 (N=1422) | Part 2: mRNA-1273 (N=1402)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (6) | 16 (17) | 12 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (5) | 4 (4)
Fatigue (General disorders) | 4 (4) | 4 (4) | 19 (19) | 10 (10)
Seasonal allergy (Immune system disorders) | 1 (1) | 3 (3) | 11 (11) | 19 (20)
Asymptomatic COVID-19 (Infections and infestations) | 2 (2) | 4 (4) | 12 (12) | 8 (8)
COVID-19 (Infections and infestations) | 28 (28) | 30 (30) | 60 (60) | 51 (51)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 26 (26) | 19 (19)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 9 (10) | 5 (5) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 8 (8) | 13 (14)
Headache (Nervous system disorders) | 6 (6) | 9 (12) | 40 (43) | 29 (29)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 4 (4) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 13 (13) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 5 (5) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 4 (4) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 22 (23) | 24 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT05249829/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT05249829/SAP_001.pdf